CLINICAL TRIAL: NCT03695211
Title: A Randomized Controlled Clinical Trial of Ultrasound-guided Superficial Cervical Plexus Block Positioned by the Great Auricular Nerve or Conventional Landmark Technique
Brief Title: Ultrasound-guided Precise Superficial Cervical Plexus Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xin Jiang, MD (Other)
Responsible Party: Sponsor-Investigator, Xin Jiang, MD, Principal Investigator, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHANGZHENG2018-19
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-04

CONDITIONS: Superficial Cervical Plexus Block
Keywords: great auricular nerve; sternocleidomastoid muscle; ultrasound guidance

STUDY DESIGN:
Intervention Model Description: Randomize, double blind, prospective
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and observers are blinded to the block position of the superficial cervical plexus
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LM group (Active Comparator): LM group use conventional landmark technique, which selects the midpoint of the posterior border of the sternocleidomastoid muscle as the puncture point of superficial cervical plexus block
  Interventions: Procedure: Conventional landmark technique
- GAN Group (Experimental): This group firstly locate the superficial cervical plexus by ultrasound scanning of the point where the great auricular nerve emerges the posterior border of the sternocleidomastoid muscle (GAN Point). GAN Group apply the precise block technique, selects the GAN Point as the puncture point of superficial cervical plexus block
  Interventions: Procedure: Precise block technique

INTERVENTIONS:
Procedure: Conventional landmark technique — inject at the midpoint of the posterior border of the sternocleidomastoid muscle
  Arms: LM group
Procedure: Precise block technique — inject at the point where the great auricular nerve emerges the posterior border of the sternocleidomastoid muscle
  Arms: GAN Group

SUMMARY:
This prospective, randomized, observer-blinded study compared ultrasound-guided superficial cervical plexus block positioned by the great auricular nerve or conventional landmark technique.

DETAILED DESCRIPTION:
Ultrasound guidance has become a reliable adjunct for brachial plexus, femoral, and sciatic nerve blocks. Furthermore, US can also be used to anesthetize purely sensory nerves such as the lateral femoral cutaneous and saphenous nerves. The superficial cervical plexus (SCP), a sensory neural plexus, supplies the skin overlying the ear, neck, angle of the mandible, shoulder, and clavicle. Traditionally, the SCP is blocked using a subcutaneous infiltration of local anesthetics along the posterior border of the sternocleidomastoid muscle. Unlike brachial plexus, sciatic nerve, etc., the SCP often cannot be displayed directly under ultrasound. The purpose of ultrasound guidance was to inject the local anesthetic solution into the correct intermuscular plane between the sternocleidomastoid and scalene muscles. In previous studies, the midpoint of the posterior border of the sternocleidomastoid muscle was often selected as the puncture point. Studies of ultrasound-guided superficial cervical plexus block are mostly unsatisfactory. Ultrasound guidance does not increase the success rate of SCP block compared with traditional technique.

The conventional landmark ultrasound guidance technique (LM group) selects the midpoint of the posterior border of the sternocleidomastoid muscle as the puncture point, but the anatomical difference of the individual cannot be considered. It may be the reason why ultrasound guidance cannot improve the success rate of the SCP block.

The great auricular nerve is the largest branch of the SCP and can be identified under ultrasound. This study intends to indirectly locate the SCP by ultrasound scanning of the point where the great auricular nerve emerges the posterior border of the sternocleidomastoid muscle (GAN Point). The method of precise SCP block at GAN Point under ultrasound guidance (GAN Group) was explored and compared with the LM Group.

ELIGIBILITY:
Inclusion Criteria:

* Patients of American Association of anesthetists（ASA）Grade 1、2 or 3
* Patients undergoing neck and shoulder surgery

Exclusion Criteria:

* Communication barriers, unable to objectively describe symptoms
* Nerve block contraindicated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of block success rate in each group | up to 15minutes
  Sensory blockade of the lesser occipital, greater auricular, transverse cervical, and supraclavicular nerves was graded according to a 3-point scale using a pinprick test: 2 = no block, 1 = analgesia (patient can feel touch, not pain), 0 = anesthesia (patient cannot feel touch). We considered a block to be successful if, at 15 mins, a score of 0 or 1 was achieved for each of the 4 nerves.

SECONDARY OUTCOMES:
Comparison of onset time of success block in each group | up to 15minutes
  onset time means time interval from completion of injection to block score of 0(patient cannot feel touch) or 1(patient can feel touch, not pain)
Comparison of pain score after surgery at PACU in each group | Day of surgery, Arrival time of PACU
  Use NRS score to assess pain level, The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. 0 means no pain, 1-3 means mild pain, 4-6 means moderate pain, 7-10 means severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Jiang, M.D, Principal Investigator — Changzheng Hospital
Locations (1):
- Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided